CLINICAL TRIAL: NCT05904613
Title: Retrospective Study Evaluating the Impact of the XEN® Implant on Endothelial Cell Density Measured Using Specular Microscopy at 3 Years After Surgery
Brief Title: Evaluation of the Impact of the XEN® Implant on Endothelial Cell Density, 3 Years After Surgery
Acronym: RETROXEN
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RETROXEN
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma
Keywords: glaucoma; Xen implant
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glaucoma is a blinding optic neuropathy affecting 80 million people worldwide, with primary open-angle glaucoma being the most common etiology. Today, the therapeutic arsenal includes drug-based hypotonizing treatments, lasers and surgery. In France, the most common surgical techniques are trabeculectomy and deep non-perforating sclerectomy (SPNP). The principle behind these filtering techniques is to lower intraocular pressure (IOP) by creating an escape route for aqueous humor from the anterior chamber (AC) of the eye into the subconjunctival space, creating a filtration bubble (FB).

A new minimally invasive treatment option has been developed to limit intra- and post-operative complications. This new technique is based on an ab interno approach, with implantation through the anterior chamber of a 6mm-long, 45µm-lumen collagen tube called XEN®. As a result, there is no dissection of the conjunctivotenone planes, as is the case in traditional surgery.

Since June 2017, surgeons have been able to use the XEN® technique in the ophthalmology department at GHPSJ.

Today, no study has yet assessed endothelial cell loss more than 2 years after this surgery. Indeed, the presence of an anterior chamber device of any type can be associated with endothelial cell loss, which increases over time well after the surgical procedure, and may require removal of the device several years after surgery.

Recent studies have investigated peripheral endothelial cell loss with other drainage systems. They show a significant decrease in peripheral endothelial cell density in relation to the implant placed in the anterior chamber. The aim of this study is to evaluate central and peripheral endothelial cell density in the long term after XEN® placement. At the visit more than 3 years after XEN® implant placement, IOP and pachymetry measurements were taken, along with a measurement of peripheral and central endothelial cell density. Corneal peripheral endothelial cell density is measured on the different quadrants of the treated eye, as well as on the controlateral eye. Measurements will be made for each eye for patients undergoing surgery on both eyes.

DETAILED DESCRIPTION:
Glaucoma is a blinding optic neuropathy affecting 80 million people worldwide, with primary open-angle glaucoma being the most common etiology. Today, the therapeutic arsenal includes drug-based hypotonizing treatments, lasers and surgery. In France, the most common surgical techniques for glaucoma are trabeculectomy and deep non-perforating sclerectomy (SPNP). These are two filtering techniques designed to lower intraocular pressure (IOP) by creating an escape route for aqueous humor from the anterior chamber (AC) of the eye into the subconjunctival space, creating a filtering bubble (FB). They can be performed alone, or at the same time as cataract surgery. The short-term complications encountered with these techniques are early hypotony and its attendant complications (choroidal detachment, hypotonic maculopathy, haemorrhages, etc.), the most frequent cause of which is conjunctival leakage of the bubble. In the medium term, tension rises with a deep anterior chamber are evidence of an over-tight scleral flap, which may require suture lysis. Finally, problems of excessive conjunctivotenone scarring affect 25% to 30% of patients, and are responsible for the majority of late tension increases. In the longer term, the most frequent complication is cataract. The rarest but most serious complication is infection of the BF, which occurs more frequently when the walls of the BF are ischemic or perforated. It can be complicated by endophthalmitis, which can lead to irreversible loss of visual acuity.

A new minimally invasive treatment option has been developed to limit intra- and post-operative complications. This new technique is based on an ab interno approach, with implantation through the anterior chamber of a 6mm-long, 45µm-lumen collagen tube called XEN®. There is no need to dissect the conjunctivotenon planes, as is the case with traditional surgery.

The geometry of the XEN® implant has been designed to prevent major hypotonia. This new technique avoids the complications associated with conjunctival dissection, while being faster and offering a standardized surgical technique. ). Today, XEN® implant placement is used in simple surgery or combined with cataract surgery for open-angle glaucoma, incipient to moderate, associated or not with a cataract, progressive and unbalanced under local hypotonizing treatment.

Since June 2017, surgeons have been able to use the XEN® technique in the GHPSJ ophthalmology department.

To date, no study has assessed endothelial cell loss more than 2 years after this surgery. Indeed, the presence of an anterior chamber device of any type may be associated with endothelial cell loss that increases over time, well after the operation, and may require removal of the device several years after the operation. One study showed that the microinvasive ab interno Alcon Cypass® device (a device similar to XEN®) caused significant endothelial cell loss 2 years after device implantation, and was unacceptable compared with conventional glaucoma surgery. The damage was proportional to the surface area of the implant in the anterior chamber, and led to the immediate withdrawal of the device from the market.

Recent studies have examined peripheral endothelial cell loss with other drainage systems. They show a significant reduction in peripheral endothelial cell density in relation to the implant placed in the anterior chamber. Intracameral devices appear to have an impact on endothelial integrity. To date, no study has assessed long-term central and peripheral endothelial cell density after XEN® placement.

At the visit more than 3 years after XEN® implantation, intraocular pressure (IOP) is measured with a Goldmann applanation tonometer, pachymetry with a NIDEK automatic refractometer and central and peripheral endothelial cell density with a NIDEK specular microscope. Peripheral corneal endothelial cell density is measured on the various ocular quadrants. The same measurements are taken on the controlateral eye. Patients undergoing surgery on both eyes receive the same measurements for each eye.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* French-speaking patient
* Patients treated for primary open-angle glaucoma, normal-pressure glaucoma, pigmentary glaucoma or secondary glaucoma in the ophthalmology department of the Paris Saint-Joseph hospital group.
* Patients who have undergone surgery with XEN® alone or in combination with cataract surgery by lens phacoemulsification, for one or both eyes.

Exclusion Criteria:

* Patient with any other associated ophthalmological disease, other than simple cataract already operated on or operated on simultaneously with XEN® application, with no intra- or postoperative complications
* History of filtering surgery prior to XEN® treatment
* Filtering surgery after XEN® treatment
* History of vitrectomy (removal of the vitreous body from the eye)
* Angle-closure glaucoma
* Uveitic glaucoma (linked to inflammation which may itself have an effect on the cornea)
* Pre-existing endothelial dystrophy, iridocorneoendothelial syndrome (ICE) (glaucoma with corneal pathology)
* Endothelial cell count below 1000 cells
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for primary open-angle glaucoma, normal-pressure glaucoma, pigmentary glaucoma or secondary glaucoma in the ophthalmology department of the Paris Saint-Joseph hospital group.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
assessment of long-term (>3years) central and peripheral endothelial cell density after XEN® placement. | at least 3 years after surgery
  Difference in central and peripheral endothelial cell density between the upper nasal quadrant and the other quadrant (lower nasal, upper and lower temporal quadrant)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France